CLINICAL TRIAL: NCT00554567
Title: Utilization of Decentralized HIV Testing and Care Services in Rural Maharashtra, India
Brief Title: Utilization of HIV Clinical Services in Rural India
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Health Management, Pachod, India (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Gita Sinha, MD MPH, Johns Hopkins University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: VCTUtilizationStudy2007
Record Dates: First submitted 2007-11-05; First posted 2007-11-07 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2008-12

CONDITIONS: HIV Infections; Sexually Transmitted Infections
Keywords: HIV/AIDS; Voluntary Counseling and Testing; Rural India; HIV Care; Health Services Research
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases; Acquired Immunodeficiency Syndrome | interventions — HIV Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention Arm (Experimental): Fully Decentralized HIV Testing and Care Services
  Interventions: Behavioral: HIV Testing and Care Services

INTERVENTIONS:
Behavioral: HIV Testing and Care Services — Fully-decentralized HIV Voluntary Counseling and Testing and referral for care

SUMMARY:
This community-based clinical trial based in two districts of rural Maharashtra, India compares utilization of an intervention model of "fully-decentralized," or rural primary clinic-based, HIV testing and care services, with a control model of the Indian government's partially-decentralized HIV services, offering rural referral clinic testing and urban-based HIV care.

DETAILED DESCRIPTION:
India has one of the highest estimated number of HIV cases globally. Sixty percent of its HIV cases occur in rural residents, yet there is no system of HIV testing or care services for them. Preliminary studies have identified very low HIV testing utilization among men and recently pregnant women in rural Maharashtra, even though these are, by government policy, high-priority target groups for rural HIV testing, diagnosis, and prevention.

This study will compare two models of rural HIV testing and care services in two districts of Maharashtra, India. The "Control" model is the Indian government's current strategy of "partially decentralized" rural-based HIV testing services at a secondary-level Community Health Center clinic, which serves a village group population of 30,000. HIV care including antiretroviral therapy is provided a the rural district headquarters in the district urban center. The "Intervention" model is a novel model of "fully decentralized" rural-based HIV testing which will be offered at the Community Health Center, two Primary Health Centers, and eight village-level sub-center clinics, and HIV care offered at a rural-based clinic.

The primary outcomes of this trial are to assess and compare utilization rates for these two types of HIV services models among rural adult men age 18-49 and pregnant women age 18 and older. Additionally, the secondary outcomes include comparing HIV clinical and behavioral risk characteristics of services utilizers in each model, and characteristics of utilizers versus non-utilizers between and within each model. Clinical care outcomes include WHO Clinical stage at time of HIV diagnosis and at first clinical care visit, and birth outcomes for HIV-infected pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Adult Male Age 18 - 49 or Pregnant Female age 18 and older
* Capacity to give written informed consent

Exclusion Criteria:

* Refusal, or Physical or Mental incapacity to give written informed consent

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1300 (Actual)
Dates: Start 2007-01; Primary Completion 2010-11 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Utilization of HIV Testing | Annual

SECONDARY OUTCOMES:
Proportion with Sexually Transmitted Infection History | Annual
Proportion with Behavioral HIV risk history | Annual
WHO Clinical Stage at time of HIV diagnosis | Quarterly
WHO Clinical Stage at first clinical care visit | Quarterly
Birth outcomes for HIV-infected pregnant women | Quarterly
Awareness of HIV Testing Services | Annual

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Dyalchand, MD MPH, Principal Investigator — Institute for Health Management, Pachod (IHMP), Maharashtra, India; Gita Sinha, MD, Principal Investigator — Johns Hopkins University School of Medicine, Baltimore, USA
Locations (1):
- Institute of Health Management, Pachod (IHMP), Pachod, Aurangabad District, Maharashtra, India

REFERENCES:
- [Result] Sinha G, Dyalchand A, Khale M, Kulkarni G, Vasudevan S, Bollinger RC. Low utilization of HIV testing during pregnancy: What are the barriers to HIV testing for women in rural India? J Acquir Immune Defic Syndr. 2008 Feb 1;47(2):248-52. PMID 18340657
- [Result] Celentano DD. Is HIV screening in the labor and delivery unit feasible and acceptable in low-income settings? PLoS Med. 2008 May 6;5(5):e107. doi: 10.1371/journal.pmed.0050107. PMID 18462015